CLINICAL TRIAL: NCT01746329
Title: Exploratory Study on the Effect of Nutritional Intervention on Postprandial Skeletal Muscle Microcirculation in Obese Subjects
Brief Title: Tea-beetroot-venous Occlusion Plethysmography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: FDS-BNH-0809; Arnhem-Nijmegen 2012/357 (Other: Commissie Mensgebonden Onderzoek)
Record Dates: First submitted 2012-11-30; First posted 2012-12-10 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Insulin Resistance; Obesity
Keywords: Obesity, insulin resistance, muscle perfusion
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tea (Experimental): Oral intake of tea containing 75 grams of glucose
  Interventions: Other: Tea
- Beet root (Experimental): Oral intake of beetroot juice containing 75 grams of glucose
  Interventions: Other: Beet root
- Placebo (Placebo Comparator): Oral intake of 75 grams of glucose in water
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Tea — Oral intake of tea containing 75 grams of glucose
  Arms: Tea
Other: Beet root — Oral intake of beetroot juice containing 75 grams of glucose
  Arms: Beet root
Other: Placebo — Oral intake of 75 grams of glucose in water
  Arms: Placebo

SUMMARY:
In the present study, muscle perfusion will be studied before and after an oral glucose challenge following a fasting period.

DETAILED DESCRIPTION:
Based on data from previous studies, this physiological response is blunted in obese subjects, and the investigators expect these responses to be restored when the glucose load is combined with tea or beetroot juice in obese, insulin resistant men.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Aged 30-70 years.
* Obesity (BMI>30 kg/m2)
* insulin resistance as fasting glucose levels >6.1 mmol/L.
* Reported intense sport activities >10 h/w.
* Reported alcohol consumption >28 units/w
* Signed Informed consent
* Currently not smoking and being a non-smoker for at least 3 months prior to the start of the study.

Exclusion Criteria:

* BMI ≥ 40 kg/m2.
* Presence of cardiovascular disease.
* Presence of sudden cardiac death in a 1st degree relative at an age <50 years.
* Presence of diabetes mellitus type 2.
* Regular tea drinker (> 2 cups per day)

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Vascular resistance | Average of values obtained at 30, 60, 90, 120, 150 and 180 minutes after test product intake corrected for the value obtained at approximately 20 minutes before test product intake (baseline)
  Vascular resistance (arm and leg) as obtained from venous occlusion plethysmography and corrected for blood pressure

SECONDARY OUTCOMES:
echo-Doppler | Approximately 20 minutes before (baseline) and 30, 60, 90, 120, 150 and 180 minutes after test product intake
  Postprandial muscle blood flow (arm and leg) measured by echo-Doppler at the brachial artery and the superficial femoral artery
Near-infrared spectroscopy | Approximately 20 minutes before (baseline) and 30, 60, 90, 120, 150 and 180 minutes after test product intake
  Postprandial muscle blood flow (arm) measured by near-infrared spectroscopy on the extensor carpi radialis brevis muscles of the forearm
Glucose and insulin | Approximately 20 minutes before (baseline) and 30, 60, 90, 120, 150 and 180 minutes after test product intake
  Glucose and insulin in venous blood plasma
Vascular resistance exploratory | Approximately 20 minutes before (baseline) and 30, 60, 90, 120, 150 and 180 minutes after test product intake
  Vascular resistance (arm and leg) as obtained from venous occlusion plethysmography and corrected for blood pressure as an exploratory parameter.

CONTACTS AND LOCATIONS:
Overall Officials: M Hopman, Prof DR, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Fuchs D, Nyakayiru J, Draijer R, Mulder TP, Hopman MT, Eijsvogels TM, Thijssen DH. Impact of flavonoid-rich black tea and beetroot juice on postprandial peripheral vascular resistance and glucose homeostasis in obese, insulin-resistant men: a randomized controlled trial. Nutr Metab (Lond). 2016 May 13;13:34. doi: 10.1186/s12986-016-0094-x. eCollection 2016. PMID 27182277